CLINICAL TRIAL: NCT01280513
Title: Influence of a Protein Diet on the Colonic Metabolism and Phosphorus Housekeeping in Healthy Volunteers.
Brief Title: Effect of Increased Protein Intake on Colonic Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor Kristin Verbeke, Ph. D., KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ML5174
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Protein Fermentation; Toxicity in the Colon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Protein intake (Experimental)
  Interventions: Dietary Supplement: High protein intake
- Low Protein intake (Experimental)
  Interventions: Dietary Supplement: Low Protein intake

INTERVENTIONS:
Dietary Supplement: High protein intake — 30% of energy intake coming from proteins
  Arms: High Protein intake
Dietary Supplement: Low Protein intake — 9% of energy intake coming from proteins
  Arms: Low Protein intake

SUMMARY:
The purpose of this study is to modulate the protein fermentation and to investigate the effect on colon toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Regular eating pattern (3 meals/day)
* Age between 18 and 45 years old
* BMI between 18,5 and 30 kg/m²

Exclusion Criteria:

* Intake of antibiotics in the last month before the study
* Abdominal surgeries in the past (accept appendectomy)
* Consulting a dietician/following a diet
* Vegetarian
* Intake of pre- and/or probiotics
* Exposure to radioactivity in the year proceeding the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Fecal water toxicity | Participants were followed for 5 weeks, with measurements on 3 specific time points

CONTACTS AND LOCATIONS:
Locations (1):
- KULeuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Windey K, De Preter V, Louat T, Schuit F, Herman J, Vansant G, Verbeke K. Modulation of protein fermentation does not affect fecal water toxicity: a randomized cross-over study in healthy subjects. PLoS One. 2012;7(12):e52387. doi: 10.1371/journal.pone.0052387. Epub 2012 Dec 20. PMID 23285019